CLINICAL TRIAL: NCT01047774
Title: Soy-rich Diet for Preventing Chronic Pain After Breast Cancer Surgery
Brief Title: The Effect of Soy Protein on Post- Breast Cancer Surgery Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty with recruitment - few eligible for enrolment.
Sponsor: Dr. Yoram Shir (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Louise & Alan Edwards Foundation (Unknown); McGill University (Other)
Responsible Party: Sponsor-Investigator, Dr. Yoram Shir, Doctor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A02-M102-07A; 5R21CA125873-02 (NIH)
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Pain; Chronic Disease; Breast Cancer
Keywords: soy protein; diet
MeSH Terms: conditions — Pain; Chronic Disease; Breast Neoplasms | interventions — Soybean Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Soy protein (Experimental)
  Interventions: Dietary Supplement: Isolated soy protein
- Milk protein (Placebo Comparator)
  Interventions: Dietary Supplement: Isolated milk protein

INTERVENTIONS:
Dietary Supplement: Isolated soy protein — 30-50g of protein powder daily for 2 weeks.
  Other Names: PRO-FAM 873; Code #066873
  Arms: Soy protein
Dietary Supplement: Isolated milk protein — 30-50g of protein powder daily for 2 weeks.
  Other Names: PRODIET 85
  Arms: Milk protein

SUMMARY:
The incidence of chronic pain after breast cancer surgery (CPBCS) is high in women diagnosed with breast cancer. Similar to other chronic postoperative pain conditions, existing treatments for CPBCS do not always work. Adopting the concept of using pain relieving measures prior to surgery rather than after it, may lead to decreased postoperative pain levels. Soy has been shown to have pain-relieving properties and may reduce the risk for developing chronic post-surgical pain. The purpose of this study is to determine the effects of adding soy protein to the diet before surgery on the development of chronic pain.

DETAILED DESCRIPTION:
Preclinical studies indicate that soy consumption suppresses the development of pain behavior and hyperalgesia following nerve injury. The pain-suppressing properties of soy protein have been shown to be predominately the result of soy pre-operative consumption.

This is a randomized, double blind, placebo-controlled clinical trial for women diagnosed with breast cancer and scheduled to undergo breast cancer surgery. The trial will comprise two phases: 1. A 2-week preoperative dietary manipulation phase, and 2. A one-year postoperative follow up period. In the first phase eligible candidates will undergo a basic dietary evaluation followed by stratification into 4 study groups, based on their pre-vs. postmenopausal status and the planned type of surgery, i.e., formal mastectomy vs. breast-conserving surgery. Women in each group will be randomized to receive either powdered soy protein in the experimental group or milk protein in the control group. During the second, post-surgical phase women will resume their normal diet. If shown to be beneficial, this simple dietary manipulation may prevent one of the most severe sequelae of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with breast cancer and scheduled for elective breast cancer surgery (excluding breast biopsy) with axillary lymph node dissection (total and/or sentinel node excision).
* Women who are 21 years or older.

Exclusion Criteria:

* History of significant heart, gastro-intestinal, liver or kidney disease.
* Use of the anticoagulant, warfarin or Coumadin.
* Malabsorption of any kind.
* Diagnosed lactase deficiency.
* Known allergy to any of the tested dietary products.
* Basic daily consumption of soy protein in quantities exceeding 10 g/day.
* Women who are strict vegetarians (i.e. no animal derived dietary sources).
* The use of the following narcotics or adjuvant pharmacotherapy: opioids, anticonvulsants, antidepressants and steroids (except antidepressant use specifically for depression).
* Tumour size (if known) > 3cm(i.e. size before pre-operative chemotherapy, if administered).
* Locally advanced breast cancer.
* Inflammatory breast cancer.
* Paget's disease of the breast with palpable mass.
* Suspected metastasis.
* Suspected micrometastasis.
* Previous breast surgery of any kind (except needle biopsy).
* The need for bilateral breast surgery.
* The existence of other known cancer, including metastasis, either in the other breast or elsewhere.
* Previous or current endocrine cancer therapy (e.g. selective estrogen receptor modulators, aromatase inhibitor).
* Body mass index (BMI) > 35.

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Number of women in both arms with any pain of any type in operated breast or its vicinity | 12 months post-surgery

SECONDARY OUTCOMES:
Pain intensity (acute) | Up to 7 days post-surgery
Pain intensity (chronic) | Up to 12 months post-surgery
Analgesic medication use | Up to 12 months post-surgery
Pain quality | Up to 12 months post-surgery
Anxiety and Depression | Up to 12 months post-surgery
Disability | Up to 12 months post-surgery
Adverse events | 2 weeks during dietary supplementation
Childhood and adolescence consumption of soy | Baseline
Adverse events | Up to 12 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Shir, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (4):
- Canada (4):
  - Royal Victoria Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - St. Mary's Hospital Center, Montreal, Quebec